CLINICAL TRIAL: NCT02720809
Title: Helbred2016: Monitorering af Kroniske Sygdomme og Risikofaktorer i Befolkningen
Brief Title: Health2016: Monitoring Chronic Disease and Risk Factors in the General Population
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Glostrup University Hospital, Copenhagen (Other)
Responsible Party: Principal Investigator, Allan Linneberg, Head of Section, Glostrup University Hospital, Copenhagen
Other Study IDs: H-15017277
Record Dates: First submitted 2016-03-22; First posted 2016-03-28 (Estimated); Last update posted 2016-03-28 (Estimated); Status verified 2016-03

CONDITIONS: Micronutrient Deficiency; Cardiovascular Disease; Allergy; Respiratory Disease
Keywords: micronutrients; blood pressure; allergy; lung function
MeSH Terms: conditions — Cardiovascular Diseases; Hypersensitivity; Respiration Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — serum, plasma, whole blood, urine
Oversight: Data Monitoring Committee: No

SUMMARY:
Health2016 is a general population cross-sectional study aimed at completing af monitoring program for monitoring chronic disease and risk factors in the period 2006 to 2016. Similar studies have been performed in 2006, 2010, and 2013.

DETAILED DESCRIPTION:
A random sample of 18-69 year-olds living in 10 municipalities in the Capital Region of Denmark is invited to a health examination including measurements of anthropometry, lifestyles, symptoms and diagnoses of diseases, blood pressure, resting heart rate, muscle strength, fitness, lung function, allergy tests, and biochemistry (lipids, liver and kidney function, vitamin D status, salt excretion, iodine status). Trends in these parameters over time will be assessed.

ELIGIBILITY:
Inclusion Criteria: General population sample randomly selected from persons living in 10 municipalities in the Capital Region of Denmark. Age 18-69 years. Danish citizenship, born in Denmark

Exclusion Criteria:

* pregnancy

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: General population sample randomly selected from persons living in 10 municipalities in the Capital Region of Denmark. Age 18-69 years.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2016-05; Primary Completion 2017-08 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
Change in micronutrient status from 2006 to 2016 | 10 years
  Serum 25-OH Vitamin D status (nmol/l) in serum from 2006 to 2016

SECONDARY OUTCOMES:
Change in HbA1C from 2006 to 2016 | 10
  Changes in HbA1C from 2006 to 2016
Change in allergic respiratory disease from 2006 to 2016 | 10 years
  Changes in prevalence of skin prick test reactivity to inhalant allergens
Change in prevalence of hypertension from 2006 to 2016 | 10 years
  Blood pressure above 140/90 or treatment for hypertension

CONTACTS AND LOCATIONS:
Overall Officials: Allan Linneberg, MD, PhD, Principal Investigator — Center for Health, The Capital Region of Denmark
Locations (1):
- Research Centre for Prevention and Health, Copenhagen, Glostrup, Denmark

IPD SHARING:
Plan to Share IPD: No